CLINICAL TRIAL: NCT03634878
Title: Evaluation of the Position of Promontofixation Prostheses in Perineal Ultrasound
Acronym: PROMONOTECHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PROMONTECHO
Record Dates: First submitted 2018-08-06; First posted 2018-08-17 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Prolapse of the Uterus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Perineal ultrasound to visualize the strips and their position (Experimental)
  Interventions: Other: perineal ultrasound

INTERVENTIONS:
Other: perineal ultrasound — Ultrasound measurement of the size and position of the prostheses.

SUMMARY:
Indirect promontofixation with prostheses is the standard surgical technique for the reference of uterine prolapse. There is no validated examination to control the position of the prostheses postoperatively.

These prostheses are echogenic and perineal ultrasound could be a means of postoperative monitoring. There is no data in the literature on the relationship between prosthesis position and postoperative symptoms

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of female sex
* Patient with double laparoscopic promontofixation without associated hysterectomy

Exclusion Criteria:

* History of hysterectomy
* Anterior cure (before index intervention) of prolapse with placement of prosthetic material.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the reproducibility study of intra and interobserver measurements of the size of promontofixation prostheses | 10 minutes
Evaluate the reproducibility study of intra and interobserver measurements position of promontofixation prostheses | 20 minutes

SECONDARY OUTCOMES:
Collect the position of the strips | 20 minutes
Collect the symptoms of the patients | 20 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Xaviar FRITEL, Principal Investigator — Poitiers University Hospital
Locations (1):
- Chu de Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: No